CLINICAL TRIAL: NCT05876299
Title: The Anabolic Properties of a Lipid-rich Pork Matrix
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 23257
Record Dates: First submitted 2023-05-16; First posted 2023-05-25 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Muscle Protein Synthesis

STUDY DESIGN:
Intervention Model Description: This study will employ a semi-crossover model whereby participants will complete 2 of 3 conditions, each.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Low-Fat Pork (Active Comparator): This condition will consist of consuming 90.2 g of low-fat (4.90% crude fat) ground pork.
  Interventions: Other: 95.1% Lean Pork
- High-Fat Pork (Experimental): This condition will consist of consuming 109.6 g of high-fat (18.84% crude fat) ground pork.
  Interventions: Other: 81.16% Lean Pork
- Carbohydrate Control (Placebo Comparator): This condition will consist of a carbohydrate beverage.
  Interventions: Other: Carbohydrate Beverage

INTERVENTIONS:
Other: 95.1% Lean Pork — This intervention will contain 120 kcals, 4.4 g fat, and 20 g protein from low-fat ground pork.
  Arms: Low-Fat Pork
Other: 81.16% Lean Pork — This intervention will contain 266 kcals, 20.6 g fat, and 20 g protein from high-fat ground pork.
  Arms: High-Fat Pork
Other: Carbohydrate Beverage — This intervention will contain 266 kcals and 73.3 g carbohydrate from a carbohydrate beverage.
  Arms: Carbohydrate Control

SUMMARY:
The amount and quality of skeletal muscle mass determines physical performance, but also a significant contributor to metabolic health. As such, the maintenance of skeletal muscle mass is relevant across the lifespan to remain active in family and community life. Food ingestion, particularly protein, is one of the main anabolic to skeletal muscle tissue by stimulating muscle protein synthesis rates. There have been multiple attempts to identify specialized performance nutrition products (e.g., various isolated protein powders) to maximize the anabolic properties of dietary protein on muscle. Our research group, however, has advocated for a food focus approach to meet dietary protein requirements. Particularly, we propose that whole foods demonstrate food matrix effects (nutrient-nutrient interactions) that creates a greater anabolic action on muscle beyond what amino acids can create alone. Therefore, the objective of this study is to identify the anabolic properties of consuming lipid-rich pork products when compared to their leaner counter-parts. Our working hypothesis that the ingestion of 84% or 96% lean ground pork condition will stimulate a greater increase in muscle protein synthesis rates compared to an isocaloric carbohydrate beverage in healthy adults. We further hypothesize that the ingestion of 84% lean pork will augment the stimulation of muscle protein synthesis rates to a greater extent than 96% lean ground pork. To achieve our objective, we will recruit 15 healthy men and women (20-50 y) to receive prime-constant infusions to directly measure muscle protein synthesis rates before and after treatment ingestion using our lab's established methods.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-50 yrs
* Pre-menopausal
* Recreationally active
* Weight stable for prior 6 months

Exclusion Criteria:

* Age outside of range (20 - 50 yrs)
* Pregnancy
* Irregular menstrual cycles
* Participation in previous research using [13C6]phenylalanine
* Participation in other ongoing research that interferes with this study (e.g., conflicting diet, activity interventions, etc.)
* Any hospitalization or surgery for a metabolic, cardiovascular, or neuromusculoskeletal complication within the past year
* Allergy or hypersensitivity to local anesthetics, latex, or adhesives (bandages, medical tape, etc.)
* Excess scarring after injury
* History of excess bleeding after cut
* Chronic or frequent dizziness/fainting, and arm or leg weakness/numbness
* Arthritis
* Tumors
* Mental Illness
* Hepatorenal, cardiovascular musculoskeletal, autoimmune, or neurological disease or disorder
* Predisposition to hypertrophic scarring or keloid formation
* Physical activity limitations
* Consumption of ergogenic-levels of dietary supplements that may affect muscle mass (e.g., creatine, HMB), insulin-like substances, or anabolic/catabolic pro-hormones (e.g., DHEA) within 6 weeks prior to participation
* Consumption of thyroid, androgenic, or other medications known to affect endocrine function
* Consumption of medications known to affect protein metabolism (e.g., prescription-strength corticosteroids, non-steroidal anti-inflammatories, or acne medication)
* Unwillingness to comply with study procedures
* Weight unstable (variation >5% of bodyweight in last 6-12 months)
* Current or previous tobacco use with last 6 months
* Obesity (body mass index; BMI > 30 kg/m^2)
* Score of less than 14 or greater than 24 on Godin-Shephard Leisure-Time Physical Activity Questionnaire
* Phenylketonuria
* Anyone hospitalized previously for COVID-19 without a cardiovascular workup screening for cardiovascular issues post-infection
* Anyone recovering from COVID-19 infection within the preceding 10 days

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2023-07-15 (Actual); Primary Completion 2024-04-09 (Actual); Study Completion 2024-04-09 (Actual)

PRIMARY OUTCOMES:
Myofibrillar Fractional Synthetic Rate | During 5-hour post-prandial period following consumption of the study meal or beverage
  Rate of building new protein in skeletal muscle contractile protein

SECONDARY OUTCOMES:
Plasma Amino Acid Concentration | During the 3-hour post-absorptive period prior to ingestion of the study meal or beverage and throughout the 5-hour post-prandial period following meal ingestion
  Concentration of amino acids in plasma as determined by LC/MS/MS
Plasma Free Fatty Acid Concentration | During the 3-hour post-absorptive period prior to ingestion of the study meal or beverage and throughout the 5-hour post-prandial period following meal ingestion
  Concentration of amino acids in plasma as determined by GC-MS
Plasma Insulin Concentration | During the 3-hour post-absorptive period prior to ingestion of the study meal or beverage and throughout the 5-hour post-prandial period following meal ingestion
  Concentration of insulin in plasma as determined by commercially-available ELISA kits
Plasma Glucose Concentration | During the 3-hour post-absorptive period prior to ingestion of the study meal or beverage and throughout the 5-hour post-prandial period following meal ingestion
  Concentration of glucose in plasma as determined by an automated biochemistry analyzer (YSI)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas A Burd, PhD, Principal Investigator — University of Illinois at Urbana-Champaign
Locations (1):
- Louise Freer Hall (University of Illinois Urbana-Champaign), Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zupancic Z, Askow AT, Barnes TM, Deutz MT, Ulanov AV, Dilger RN, Dilger AC, Willard JW, Mackenzie RW, Harseim JE, Hernandez-Saavedra D, Burd NA. Ingestion of a lipid-rich meat matrix blunts the postexercise increase of myofibrillar protein synthesis rates in healthy adults: a randomized controlled trial. Am J Clin Nutr. 2025 Nov;122(5):1252-1264. doi: 10.1016/j.ajcnut.2025.09.001. Epub 2025 Sep 7. PMID 40925524